CLINICAL TRIAL: NCT03762993
Title: Vocal Restoration Programs After Acute Vocal Exertion
Brief Title: Controlled Phonation and Vocal Rest Programs After Acute Vocal Exertion in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Preeti M. Sivasankar, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Vocal restoration programs
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Within Subject Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Adults (Experimental): Participants will complete vocal rest and controlled phonation
  Interventions: Behavioral: Vocal rest and Controlled Phonation
- Healthy Adults reporting Vocal Fatigue (Experimental): Participants will complete vocal rest and controlled phonation
  Interventions: Behavioral: Vocal rest and Controlled Phonation

INTERVENTIONS:
Behavioral: Vocal rest and Controlled Phonation — Voice rest and semi occluded vocal tract voice exercises

SUMMARY:
The proposed research will investigate the most effective strategy to reduce vocal exertion reported by speakers in noisy environments. Repeated vocal exertion can lead to voice problems and therefore identifying effective strategies can lead to better prevention of acquired voice disorders. This study will compare the effects of vocal rest and controlled phonation both before and after vocal exertion. The investigators hypothesize that vocal rest and controlled phonation will mitigate the negative effects of vocal exertion.

ELIGIBILITY:
Inclusion Criteria:

* within age range

Exclusion Criteria:

* Voice Disorders
* Strong gag reflex
* Craniofacial disorders
* Cognitive Impairments
* Head and Neck Cancer
* Hearing Difficulties
* Dentition problems that prevent an oral scope being placed in mouth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Sivasankar, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 37 enrolled participants, 31 were assigned to study groups based on self-reported vocal fatigue level.
Period: Overall Study
Arm/Group | Healthy Adults | Healthy Adults Reporting Vocal Fatigue
Started | 21 | 10
Completed | 21 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Adults | Healthy Adults Reporting Vocal Fatigue | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 17 | 6 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 9 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 15 | 6 | 21
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 10 | 31
Vocal Fatigue Index [Median (Full Range); unit: units on a scale] — The Vocal Fatigue Index measures self-reported vocal fatigue symptoms. The scale is divided into three separately scored sections (two of which were used here). Possible scores range from 0 to 44 on Part 1, and 0 - 20 on part 2. Scores >24 on part 1, or >7 on part 2 are indicative of vocal fatigue.Scores below this range are considered normal.
  units on a scale
    Vocal Fatigue Index Part 1 | 4 [0 to 23] | 24 [4 to 27] | 4 [0 to 27]
    Vocal Fatigue Index Part 2 | 0 [0 to 5] | 3.5 [2 to 9] | 2 [0 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Phonation Threshold Pressure
Description: Minimum air pressure required to initiate and sustain vocal fold oscillation
Time Frame: 2.5 hours
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Healthy Adults | Healthy Adults Reporting Vocal Fatigue
Number analyzed (Participants) | 21 | 10
cmH20
  Pre-Exertion | 5.41 (1.26) | 5.08 (1.59)
  Post-Exertion | 6.39 (1.8) | 6.33 (1.4)
  Post Restoration Strategy | 5.63 (1.32) | 5.61 (1.59)
Statistical Analysis 1: Comparison: Healthy Adults vs Healthy Adults Reporting Vocal Fatigue; Test type: Other — Changes in phonation threshold pressure were analyzed using a linear mixed effect model. Fixed factors included in the statistical model included time, group, and restoration strategy (controlled phonation or vocal rest). In addition, appropriate interactions were included and participant was added as a random factor in order to control for individual variation; p < 0.001, Mixed Models Analysis — P-value is for the effect of time. A priori significance level set at .05

2. Secondary Outcome: Lung Volume Excursion
Description: The difference between lung volume initiation and termination on connected speech
Time Frame: 2.5 hours
Measure: Mean (Standard Deviation); unit: % Vital Capacity
Arm/Group | Healthy Adults | Healthy Adults Reporting Vocal Fatigue
Number analyzed (Participants) | 21 | 10
% Vital Capacity
  Baseline | 13.5 (7.2) | 14.5 (6.4)
  Post Exertion | 21.6 (10.6) | 12.9 (6.5)
  Post Restoration Strategy | 18.7 (11.5) | 18.4 (7.15)
Statistical Analysis 1: Comparison: Healthy Adults vs Healthy Adults Reporting Vocal Fatigue; Test type: Other — Changes in lung volumes were analyzed using a linear mixed effect model. Fixed factors included in the statistical model included time, group, and restoration strategy (controlled phonation or vocal rest). In addition, appropriate interactions were included and participant was added as a random factor in order to control for individual variation; p < 0.01, Mixed Models Analysis — P-value represents effect of group. A priori threshold for significance set at .05

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events from the time consent was obtained until approximately 24 hours following study completion.
Arm/Group | Healthy Adults | Healthy Adults Reporting Vocal Fatigue
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/10
Other Adverse Events (participants affected / at risk) | 0/21 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT03762993/Prot_SAP_000.pdf